CLINICAL TRIAL: NCT01032798
Title: Efficacy and Pharmacokinetics of Liposomal Mepivacaine Formulations in Dentistry
Brief Title: Local Anesthetics New Formulations: From Development to Clinical Tests
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Dr. Giovana R. Tofoli, UNICAMP
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 06/00121-9
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2007-04

CONDITIONS: Local Anesthetic Effectiveness
MeSH Terms: interventions — Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: mepivacaine — One intra-oral injection at four different sessions, of the following formulations: 2% mepivacaine with 1:100,000 epinephrine, 3% mepivacaine, 2% and 3% liposome-encapsulated mepivacaine.

SUMMARY:
This blinded cross-over study aim to evaluate the efficacy and the pharmacokinetics of a previously reported liposome-encapsulated mepivacaine formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Volunteers were free from cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and haematological diseases, psychiatric disorders and allergy to local anesthetics

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Latency period and duration of anesthesia were assessed by an electrical pulp tester | 10 minutes

SECONDARY OUTCOMES:
Plasma concentrations of mepivacaine | 0 to 360 minutes after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Eneida de Paula, PHD, Study Director — University of Campinas, Brazil
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Tofoli GR, Cereda CM, Groppo FC, Volpato MC, Franz-Montan M, Ranali J, de Araujo DR, de Paula E. Efficacy of liposome-encapsulated mepivacaine for infiltrative anesthesia in volunteers. J Liposome Res. 2011 Mar;21(1):88-94. doi: 10.3109/08982104.2010.483596. Epub 2010 May 20. PMID 20482446